CLINICAL TRIAL: NCT07348679
Title: A Randomized Trial of Charcoal-filtered Cigarettes on Product Perceptions, Smoking Behaviors, and Toxicant Exposure
Brief Title: Cigarette Filter Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa Mercincavage, PhD, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2025000854; R37CA296976 (NIH)
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Smoking ( Cigarette)
Keywords: smoking behavior; charcoal; cigarette filter; perceptions; biomarkers
MeSH Terms: conditions — Cigarette Smoking; Smoking; Anthrax | interventions — Marketing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NAS Sky charcoal-filtered cigarettes (Experimental): Charcoal-filtered cigarettes
  Interventions: Behavioral: Charcoal filtered cigarettes with marketing
- NAS Yellow non-charcoal-filtered cigarettes (Active Comparator): Conventional-filtered cigarettes
  Interventions: Behavioral: Non-charcoal filtered cigarettes
- Tareyton charcoal cigarettes (Experimental): Charcoal-filtered cigarettes
  Interventions: Behavioral: Charcoal filtered cigarette without marketing

INTERVENTIONS:
Behavioral: Charcoal filtered cigarettes with marketing — After completing a 7-day baseline period of smoking their own preferred brand, participants randomized to the charcoal filtered cigarette with marketing condition will use Natural American Spirit Sky cigarettes for the next 28 days
  Arms: NAS Sky charcoal-filtered cigarettes
Behavioral: Charcoal filtered cigarette without marketing — After completing a 7-day baseline period of smoking their own preferred brand, participants randomized to the charcoal filtered cigarette without marketing condition will use Tareyton cigarettes for the next 28 days
  Arms: Tareyton charcoal cigarettes
Behavioral: Non-charcoal filtered cigarettes — After completing a 7-day baseline period of smoking their own preferred brand, participants randomized to the non-charcoal filtered cigarette condition will use Natural American Spirit Yellow cigarettes for the next 28 days
  Arms: NAS Yellow non-charcoal-filtered cigarettes

SUMMARY:
The overall purpose of this study is to determine the effects of using charcoal-filtered cigarettes on product perceptions, smoking behaviors, and biomarkers of exposure to tobacco-related toxicants. The main questions it aims to answer are:

Do perceptions of cigarettes differ by their filter? Do people smoke charcoal-filtered cigarettes differently than cigarettes with conventional filters, and does this change their exposure to cigarette harms?

Study participants will complete a 5-week laboratory-based, open-label, parallel-design randomized trial. After a baseline period of smoking their preferred brand, participants will smoke charcoal-filtered or non-charcoal-filtered cigarettes for 4 weeks while completing weekly sessions to assess primary outcomes. During weekly sessions, they will smoke two cigarettes in our laboratory, provide urine and carbon monoxide samples, and complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be:

  1. Male and female smokers who are at least 21 years of age and self-report smoking at least 5 cigarettes per day for at least the past 6 months.
  2. Smokers of primarily non-menthol cigarettes of brands other than Natural American Spirit.
  3. Not currently undergoing smoking cessation treatment or trying to quit.
  4. Able to communicate fluently in English (speaking, writing, and reading).
  5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

* Subjects who self-report and/or present with the following criteria will not be eligible to participate in the study:

Smoking Behavior

1. Use of menthol or Natural American Spirit cigarettes as preferred/regular brand (defined as using >20% of the time).
2. Enrollment or plans to enroll in a smoking cessation program in the next month.
3. Provide an initial Carbon Monoxide (CO) reading < 5 parts per million (ppm).

Alcohol/Drugs

1. History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse.
2. Current alcohol consumption that exceeds 25 standard drinks/week.

Medical

1. Women who are pregnant, planning a pregnancy, and/or lactating.
2. Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the completion of procedures included within this protocol. Notable impairments will be evaluated by the PI and eligibility will be determined on a case-by-case basis.
3. Color blindness.
4. Serious or unstable disease within the past 12 months (e.g. heart disease, cancer). Applicable conditions will be evaluated by the Principal Investigator and eligibility will be determined on a case-by-case basis.

Psychiatric

As determined by self-report:

1. Lifetime history or current diagnosis of psychosis, bipolar disorder, and/or schizophrenia.
2. Current diagnosis of major depression. Subjects with a history of major depression, in remission for 6 months or longer, are considered eligible.

Other

Additionally, participants may be deemed ineligible for any of the following general reasons at any point throughout the study, as well as during the initial telephone screen, at the discretion of the PI:

* Significant non-compliance with protocol and/or study design.
* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact study data.
* Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk beliefs | Day 35
  Risk beliefs will be captured via 8 items rated on a 5-point Likert scale (1 = "definitely untrue", 5 = "definitely true") that evaluate participants' preferred brand and the cigarettes they smoke on the following beliefs: a) "lower in nicotine", b) "lower in tar", c) "less addictive", d) "less likely to cause cancer", e) "has fewer chemicals", f) "is healthier", g) "makes smoking safer", h) "helps people quit smoking." Individual items will be scores as correct or incorrect, and incorrect responses will be summed to created an overall false beliefs score (0-8 range, with higher scores indicating greater false beliefs about reduced risk.
Perceived health risks | Day 35
  Participants will indicate on a 7-point Likert scale (1 = "very low risk", 7 = "very high risk") their risk of developing smoking-related health conditions (i.e., lung cancer, heart disease, stroke, emphysema, respiratory infections, and other cancers) from regular use of the cigarette they are smoking. Higher mean scores indicate greater perceived risk (range 1-7).
Subjective ratings | Day 35
  Participants will rate cigarettes smoked during in-person visits using 14 individual items assessing various cigarette characteristics (e.g., strength, taste, satisfaction, harshness) used by the tobacco industry and our laboratory. Items are rated on a 100 mm visual analog scale with item-specific anchors (e.g., strength: 0 = "very weak," 100 = "very strong"); lower scores indicate less favorable ratings. We will examine mean composite scales generated from these items to assess domains of product harshness, smoking satisfaction, positive sensory experience, and cleanliness.
Daily cigarette consumption | Day 35
  Daily cigarette consumption will be assessed by participant self-report and verified through collection of used filters for all cigarettes smoked during the 5-week study. The mean will be computed for daily cigarette consumption during the week preceding final study session (i.e., mean of cigarettes smoked per day between Sessions 5 and 6, or Days 28-35).
Smoking topography (puffs taken) | Day 35
  We will use a validated procedure to score video recorded smoking sessions to quantify puffing behavior to obtain estimated number of puffs taken.
Smoking topography (total duration) | Day 35
  We will use a validated procedure to score video recorded smoking sessions to quantify puffing behavior to obtain estimates of the duration of each puff, and sum these to create a summary composite measure (in sec).
Smoking topography (total interpuff interval) | Day 35
  We will use a validated procedure to score video recorded smoking sessions to quantify puffing behavior to obtain estimates of interpuff interval (i.e., time between puffs) and created a summed composite (in sec).
Session onset carbon monoxide (CO) | Day 35
  CO will be assessed in ppm using the coVita Micro+ pro Smokerlyzer breath CO monitor (Santa Barbara, CA) at session onset to estimate daily tobacco exposure.
Carbon monoxide (CO) boost | Day 35
  CO will be assessed in ppm using the coVita Micro+ pro Smokerlyzer breath CO monitor (Santa Barbara, CA) before and after each cigarette smoked. The change in CO resulting from smoking a cigarette, CO boost, estimates exposure due to smoking an individual cigarette.
Tobacco/nicotine exposure | Day 35
  Total nicotine equivalents exposure will be assessed via measuring urine concentrations of nicotine metabolites by liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS) using Waters Xevo® TQ-XS Tandem Mass Spectrometer with ACQUITY UPLC I-Class Chromatography System (UPLC-MS-MS). Greater values indicate greater exposure.
NNAL exposure | Day 35
  We will assess NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol), a metabolite of NNK (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone), a potent lung carcinogen. A highly sensitive UHPLC-MS/MS method with Waters Xevo® TQ-XS UPLC-MS-MS will determine total NNAL in urine using liquid-liquid extraction followed by conversion to the hexanoate ester derivative. Greater values indicate greater exposure.
VOC exposure | Day 35
  We will collect a urine sample to assess exposure to seven volatile organic compounds (VOCs) due to their association with adverse health effects such as cancer, birth defects, and neurological damage S-(3-hydroxypropyl)-mercapturic acid (3HPMA, a metabolite of potentially toxic acrolein; 2-Carbamoyl-2-hydroxy-ethyl mercapturic acid (2CAHEMA, a metabolite of a neurotoxicant acrylamide); 2-carbamoyl-2-hydroxy-ethyl mercapturic acid (2CYEMA, a metabolite of a potent respiratory irritant acrylonitrile); phenyl mercapturic acid (PHMA, a metabolite of IARC Group 1 carcinogen benzene); benzyl mercapturic acid (BZMA, a metabolite of IARC Group 3 carcinogen toluene); 2,4-Dimethylphenyl mercapturic acid (24MPHMA, a metabolite of IARC Group 3 carcinogen xylene); and N-Acetyl-S-(4-hydroxy-2- buten-1-yl)-L-cysteine (MHBMA3, a metabolite of 1,3-Butadiene).

SECONDARY OUTCOMES:
End of study interview | Day 35
  We will conduct in-depth interviews with participants to qualitatively assess their reactions to the cigarettes they used during the experimental period to provide important contextual information to interpret the behavioral and survey outcome results. An interviewer will be trained with and will use an interview guide that includes open-ended questions pertaining to subjective ratings, appeal, and harm perceptions of the different types of cigarettes used in the study, with probes to inquire about associations of specific features (i.e., the charcoal filter) with reduced harm. We will also ask participants about the role of charcoal in other non-tobacco products.
Craving | Day 35
  Craving will be assessed using at session onset using the Questionnaire on Smoking Urges with a "right now" frame of reference to determine a summary score from a 32-item Likert-format self-report instrument; mean scores range from 1-7 with greater scores indicating greater craving.
Withdrawal | Day 35
  The 21-item Withdrawal Symptom Checklist (WSC) using a "right now" frame of reference, will ask participants to rate the intensity of their symptoms (e.g., cravings, irritability, difficulty concentrating) on a 4-point scale (0 = not present, 3 = severe) at session onset.
Attitudes | Day 35
  Attitudes toward study-supplied cigarettes will be assessed by the mean of an eight-item, seven-point semantic differential scale (Strasser, Cappella, et al., 2009; Yzer et al., 2003) that asks, "Which of the words below would best describe your continued use of this product?" Items were a) bad/good, b) unenjoyable/enjoyable, c) unpleasant/pleasant, d) foolish/wise, e) difficult/easy, f) more/less harmful, g) not under/under my control, and h) less/more healthy. Higher scores indicate more favorable attitudes.
Intentions | Day 35
  Two Likert-type items will assess participants' intentions to purchase and regularly use the study-supplied cigarettes, using a 5-point response scale, with greater scores indicating greater intention.
Cigarette purchase task | Day 35
  Behavioral economic indices of demand will be measured using a hypothetical purchase task that asks participants how many study cigarettes they would purchase a day at free price and across a price range guided by our previous work and a scoping review on tobacco demand.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mercincavage, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Institute for Nicotine and Tobacco Studies, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw and deidentified and recoded survey, smoking behavior, biomarker, and interview data will be preserved and shared. Respondent identifiers will not be shared. Raw audio recordings of qualitative interviews and video recordings of smoking sessions will not be shared as these cannot be fully deidentified (e.g., video recordings contain full facial images of participants); however, data derived from these recordings will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: IPD and supporting information will be made accessible as soon as possible, and no later than at the time of publication or at the end of the award, whichever comes first. Study data deposited in NAHDAP will be available to the research community in perpetuity.
Access Criteria: Deidentified study data will be made available open access without restrictions to the research community via the National Addiction & HIV Data Archive (NAHDAP). Individuals wishing to access the data must register with NAHDAP and agree to the Terms of Use, which are designed to protect the participants in the sample by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify participants, and requiring immediate reporting of any disclosure of participant identity. Data users also agree not to share or redistribute any data downloads.